CLINICAL TRIAL: NCT03758625
Title: A Phase I Study to Evaluate the Safety, Tolerability and Immunogenicity of a Therapeutic HIV Vaccine Composed of Autologous Dendritic Cells Loaded With Autologous Inactivated Whole Virus or Conserved Peptides in ART-treated HIV-infected Adults
Brief Title: Comparison of Dendritic Cell-Based Therapeutic Vaccine Strategies for HIV Functional Cure
Acronym: DC-HIV04
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sharon Riddler (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Sharon Riddler, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIDS-ES 38541; U01AI131285 (NIH)
Record Dates: First submitted 2018-11-20; First posted 2018-11-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: HIV Infections
Keywords: dendritic cell; vaccine; immunogenicity; HIV; vaccination; immune system
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, multi-arm
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- ARM A (Experimental): a1DC + inactivated whole autologous HIV vaccine given as six monthly doses of approximately 10e7 DC per dose
  Interventions: Biological: a1DC + inactivated whole autologous HIV
- ARM B (Experimental): a1DC + conserved HIV peptides vaccine given as six monthly doses of approximately 10e7 DC per dose
  Interventions: Biological: a1DC + conserved HIV peptides
- ARM C (Active Comparator): a1DC + no antigen vaccine given as six monthly doses of approximately 10e7 DC per dose
  Interventions: Biological: a1DC + no antigen
- ARM D (Experimental): pgDC + inactivated whole autologous HIV vaccine given as six monthly doses of approximately 10e7 DC per dose
  Interventions: Biological: pgDC + inactivated whole autologous HIV
- ARM E (Experimental): pgDC + conserved HIV peptides vaccine given as six monthly doses of approximately 10e7 DC per dose
  Interventions: Biological: pgDC + conserved HIV peptides
- ARM F (Active Comparator): pgDC + no antigen vaccine given as six monthly doses of approximately 10e7 DC per dose
  Interventions: Biological: pgDC + no antigen

INTERVENTIONS:
Biological: a1DC + inactivated whole autologous HIV — Investigational vaccine composed of autologous dendritic cells matured with an optimized cocktail (a1DC) and loaded with autologous -inactivated HIV
  Arms: ARM A
Biological: a1DC + conserved HIV peptides — Investigational vaccine composed of autologous dendritic cells matured with an optimized cocktail (a1DC) and loaded with a conserved HIV gag and pol peptide pool
  Arms: ARM B
Biological: a1DC + no antigen — Control vaccine composed of autologous dendritic cells matured with an optimized cocktail (a1DC) but without an antigen
  Arms: ARM C
Biological: pgDC + inactivated whole autologous HIV — Investigational vaccine composed of autologous dendritic cells matured with a standard prostaglandin E2 cocktail (pgDC) and loaded with autologous -inactivated HIV
  Arms: ARM D
Biological: pgDC + conserved HIV peptides — Investigational vaccine composed of autologous dendritic cells matured with a standard prostaglandin E2 cocktail (pgDC) and loaded with a conserved HIV gag and pol peptide pool
  Arms: ARM E
Biological: pgDC + no antigen — Control vaccine composed of autologous dendritic cells matured with a standard prostaglandin E2 cocktail (pgDC) but without an antigen
  Arms: ARM F

SUMMARY:
This study will be done in people living with HIV to see if an investigational vaccine made from a person's own white blood cells is safe and tolerated. This study will also look at the body's immune response to the vaccine and evaluate four different methods of making the vaccine to see which method may result in better immune responses.

DETAILED DESCRIPTION:
Despite the availability of strong medicines for HIV infection, there is no cure for the infection. The current anti-HIV drugs, used in combination, are effective in slowing the growth of the virus and delaying the progression of the infection. There is increasing information to suggest that a vigorous immune response (a strong response of the body to fight infection) to HIV may also result in improved control of the HIV infection. Such strong immune responses are found in a small number of HIV-infected individuals, but not in the majority.

Dendritic cells, or DCs, are a type of white blood cell that works together with other immune cells to fight infection. The DCs role is to bring substances foreign to the body, such as viruses including HIV or cancer cell proteins, to the body's immune system. Large numbers of DCs can be made from blood samples and administered back to the same person as an individualized vaccine. Vaccines made from DCs have been studied in HIV and numerous types of cancer.

The vaccines will be created by two different laboratory methods, standard or improved, using an individual's own DCs and either an individual's own inactive HIV that has been killed with heat or manmade HIV proteins called peptides. The peptides have not been studied for this use in humans, and these vaccines are not approved by the Food and Drug Administration (FDA) to prevent or treat HIV infection.

This study will be done in two steps. During Step 1 (Entry-Week 12), participants will have 4 study visits for tests, procedures and exams. At Week 4, participants will be randomized by chance into one of six study groups, like rolling dice. Four of the study groups will receive a DC-HIV vaccine while two of the study groups will receive a "control" vaccine with only DCs. Participants will have a 4:1 chance of receiving a DC-HIV study vaccine.

* Group 1: enhanced DC-HIV vaccine with inactive HIV
* Group 2: enhanced DC-HIV vaccine with HIV peptides
* Group 3: enhanced DCs only (control)
* Group 4: classic DC-HIV vaccine with inactive HIV
* Group 5: classic DC-HIV vaccine with HIV peptides
* Group 6: classic DCs only (control)

Each participant will receive 6 study vaccinations at 4-week intervals beginning at Week 12. Researchers will compare the results from participants who get the active study vaccines with results from participants who get the control vaccines. Participants, the researchers and the clinic staff will not know which vaccine participants are getting.

In Step 2 (Weeks 12 - 80), participants will have 18 study visits to receive the 6 study vaccinations and for tests to monitor health and safety and to see how the study vaccine affects the immune system and the virus.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection, documented by any FDA-approved assay. NOTE: The term 'licensed' refers to a US FDA approved kit, which is required for all investigational new drug (IND) studies.
2. Receiving continuous ART for at least 24 months (defined as no interruptions longer than 14 consecutive days) and with no changes in the components of the ART for at least 8 weeks prior to study entry. A change in formulation (for example tenofovir disaproxil fumarate to tenofovir alafenamide) will not be considered a change in ART.
3. Screening CD4+ cell count ≥350cells/mm3 obtained within 60 days prior to study entry by any US laboratory that has a CLIA certification or its equivalent.
4. Plasma HIV-1 RNA levels < 50 copies/ml for at least 24 months prior to study entry using a FDA-approved assay performed by any laboratory that has a CLIA certification or its equivalent. Participants must have at least one documented HIV-1 RNA less than 50 copies/ml >24 months prior to study entry and at least one HIV-1 RNA less than 50 copies/ml within 12 months prior to study entry. All available HIV-1 RNA measurements must be < 50 copies/ml during the 24 months prior to study entry except as allowed by the following note.

   NOTE: Unconfirmed plasma HIV-1 RNA > 50 copies/ml but <200 copies/mL is allowed if followed by a subsequent value < 50 copies/ml.
5. Screening HIV-1 RNA levels <50 copies/mL using a FDA-approved assay performed by any laboratory that has a CLIA certification or its equivalent within 60 days prior to entry.
6. Men and women age 18 to 70 years, inclusive.
7. The following laboratory values obtained within 60 days prior to entry:

   Hemoglobin ≥10 g/dL Absolute neutrophil count (ANC) ≥1000/mm3 Platelet count ≥100,000/mm3 Creatinine ≤ 1.5x upper limit of normal (ULN) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) (SGPT) ≤2.5x ULN
8. Ability and willingness of participant to provide informed consent.
9. In the opinion of the investigator, no medical, mental health or other condition that precludes participation.
10. For females of reproductive potential, negative serum or urine pregnancy test within 48 hours prior to entry by any US clinic or laboratory that has a CLIA certification or its equivalent, or is using a point-of-care (POC)/ CLIA-waived test. Females of reproductive potential include women who have not been post-menopausal for at least 12 consecutive months, (i.e., who have had menses within the preceding 12 months) or women who have not undergone surgical sterilization (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation or salpingectomy). Self- report is acceptable documentation of menopause and sterilization.
11. All participants must agree not to participate in the conception process (eg, active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, the participant/partner must use at least one reliable form of contraception (condoms, with or without a spermicidal agent; a diaphragm or cervical cap with spermicide; an IUD; or hormone-based contraceptive), while receiving study treatment and for 12 weeks following the final study vaccine.

Exclusion Criteria:

1. Currently breastfeeding or pregnant
2. Known allergy/sensitivity or any hypersensitivity to components of study vaccine or their formulation.
3. Known chronic inflammatory conditions such as, but not limited to, rheumatoid arthritis, systemic lupus erythematosus, sarcoidosis, inflammatory bowel disease (i.e., Crohn's disease or ulcerative colitis), chronic pancreatitis, or autoimmune hepatitis, myositis, or myopathy.
4. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
5. Serious medical illness that requires systemic treatment and/or hospitalization within 30 days prior to entry.
6. Use of systemic immunomodulators (eg, interleukins, interferons, cyclosporine), systemic cytotoxic chemotherapy, or investigational therapy within 60 days prior to study entry.

   NOTE: Participants receiving stable physiologic doses of glucocorticoids, defined as the equivalent of prednisone ≤10 mg/day, will not be excluded. Stable physiologic glucocorticoid doses should not be discontinued for the duration of the study. In addition, participants receiving inhaled or topical corticosteroids, or topical imiquimod will not be excluded.
7. Participation on any HIV immunotherapy or therapeutic vaccination trials within 6 months prior to study entry.
8. History of positive HCV antibody with detectable HCV RNA in plasma within 48 weeks prior to study entry.

   NOTE: Persons with positive HCV Ab but negative plasma HCV RNA are allowed to participate. Sites must document negative HCV RNA within 24 weeks of study entry.
9. History of positive HBsAg within 48 weeks prior to study entry.
10. Treatment for hepatitis C within 6 months prior to study entry.
11. Initiation of ART during acute HIV-1 infection (as determined by the site investigator by history and/or available medical records).
12. Lack of adequate venous access that, in the opinion of the investigator, would interfere with study requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of six immunizations (10e7 DCs per dose) of DC-whole virus and DC-peptide vaccines in HIV-1 infected participants on effective ART | Step 2-Week 0 (overall Study Week 12) to overall Study Week 80
  Occurrence of Grade ≥ 3 AE including signs/symptoms, lab toxicities, and/or clinical events that are possibly, probably, or definitely related to study treatment (as judged by the site investigator, blinded to treatment arm) at any time from the initial dose of DC vaccine product to end of study follow-up.
Efficacy of six immunizations (10e7 DCs per dose) of DC-whole virus and DC-peptide vaccines in HIV-1 infected participants on effective ART | Baseline to Step 2-Week 22 (overall Study Week 34)
  Change in HIV-specific CD8 and T-cell immune response as measured by ELISPOT between the vaccine arms.

SECONDARY OUTCOMES:
Relative efficacy of the DC-HIV vaccines in priming HIV-specific-CD8+ T cells | Baseline to Step 2-Week 22 (overall Study Week 34)
  Change in the ability of the DC-HIV vaccines to inhibit autologous HIV in an ex vivo virus inhibition assay.
Effect of DC-HIV vaccination on the level of persistent viremia in plasma | Baseline to Step 2-Week 22 (overall Study Week 34)
  Change in plasma HIV-1 RNA viral load as measured by single copy assay (SCA)
Effect of DC-HIV vaccination on HIV specific CD8 T-cell polyfunctional responses | Baseline to Step 2-Week 22 (overall Study Week 34)
  Change in HIV specific CD8 T-cell polyfunctional responses as measured by intracellular cytokine staining using flow cytometry.
Assess the impact of DC-HIV vaccination on levels of cell-associated HIV-1 RNA and DNA | Baseline to Step 2-Week 22 (overall Study Week 34)
  Changes in cell-associated HIV-1 RNA and DNA levels and assessment of the differences between the vaccine arms
Effect of DC-HIV vaccination on the levels of immune activation | Baseline to Step 2-Week 22 (overall Study Week 34)
  Changes in markers of cellular immune cell activation and assessment of the differences between the vaccine arms
Effect of DC-HIV vaccination on the levels of systemic inflammation | Baseline to Step 2-Week 22 (overall Study Week 34)
  Changes in soluble markers of systemic inflammation and assessment of the differences between the vaccine arms

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Riddler, MD, Study Chair — University of Pittsburgh; Bernard Macatangay, MD, Study Chair — University of Pittsburgh; John Mellors, MD, Study Chair — University of Pittsburgh
Locations (2):
- United States (2):
  - AIDS Clinical Trials Unit/The Ohio State University, Columbus, Ohio
  - HIV/AIDS Clinical Research Unit / University of Pittsburgh, Pittsburgh, Pennsylvania